CLINICAL TRIAL: NCT01010906
Title: An Open-label, 3-Part, Single-Dose Study to Investigate the Influence of Hepatic Insufficiency on the Pharmacokinetics of MK-7009
Brief Title: A Study Investigating the Influence of Hepatic Insufficiency on the Pharmacokinetics of Vaniprevir (MK-7009-005)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7009-005; 2009_674
Record Dates: First submitted 2009-11-06; First posted 2009-11-10 (Estimated); Results first posted 2014-09-29 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-09

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — vaniprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Mild Hepatic Insufficiency (HI) (Experimental): Participants with mild hepatic insufficiency (HI) administered a single 300 mg oral tablet of vaniprevir
  Interventions: Drug: Vaniprevir 300 mg
- Healthy Control to Mild HI (Experimental): Healthy, matched to mild HI, control participants administered a single 300 mg oral tablet of vaniprevir
  Interventions: Drug: Vaniprevir 300 mg
- Moderate HI (Experimental): Participants with moderate HI administered a single 300 mg oral tablet of vaniprevir
  Interventions: Drug: Vaniprevir 300 mg
- Healthy Control to Moderate HI (Experimental): Healthy, matched to moderate HI, control participants administered a single 300 mg oral tablet of vaniprevir
  Interventions: Drug: Vaniprevir 300 mg
- Severe HI (Experimental): Participants with severe HI administered a single 200 mg oral tablet of vaniprevir
  Interventions: Drug: Vaniprevir 200 mg
- Healthy Control to Severe HI (Experimental): Healthy, matched to severe HI, control participants administered a single 200 mg oral tablet of vaniprevir
  Interventions: Drug: Vaniprevir 200 mg

INTERVENTIONS:
Drug: Vaniprevir 300 mg — single dose administration of 300 mg oral tablet
  Other Names: MK-7009
  Arms: Healthy Control to Mild HI; Healthy Control to Moderate HI; Mild Hepatic Insufficiency (HI); Moderate HI
Drug: Vaniprevir 200 mg — single dose administration of 200 mg oral tablet
  Other Names: MK-7009
  Arms: Healthy Control to Severe HI; Severe HI

SUMMARY:
This was a 3-part study comparing the pharmacokinetics after administration of vaniprevir (MK-7009) for participants with mild, moderate or severe hepatic insufficiency with healthy matched control participants. The primary hypothesis is that the area under the curve (AUC) (0 to infinity) of vaniprevir for participants with mild, moderate, or severe hepatic insufficiency is similar to that observed in healthy matched controlled participants.

ELIGIBILITY:
Inclusion Criteria:

Hepatic Participants:

* Females of reproductive potential test negative for pregnancy and agree to use an appropriate method of contraception during the study
* Apart from hepatic insufficiency, is in good general health
* Has a diagnosis of chronic stable hepatic insufficiency
* Score on the Child-Pugh scale ranged from 5 to 6 (mild hepatic insufficiency); from 7 to 9 (moderate hepatic insufficiency); from 10 to 15 (severe hepatic insufficiency). Moderate and Severe participants must have had a 50% score of 2 or higher on at least one of the laboratory parameters (i.e., albumin, prothrombin time, bilirubin) at the prestudy visit.

Healthy Matched Participants:

* Females of reproductive potential test negative for pregnancy and agree to use an appropriate method of contraception during the study
* Is in good health

Exclusion Criteria:

* Female is pregnant, lactating, expecting to become pregnant or donate eggs
* Has a history of stroke or seizures
* Has a history of cancer
* Is unable to refrain from the use of any prescription or non-prescription medication
* Consumes excessive amounts of alcohol or caffeinated beverages daily
* Has had surgery, donated blood or participated in another investigational study with in the last 4 weeks
* Is a regular user or past abuser of any illicit drug including alcohol

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-07-01 (Actual); Primary Completion 2010-06-11 (Actual); Study Completion 2010-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=7009-005&kw=7009-005&tab=access

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Control for Mild HI; Healthy Control for Moderate HI: Healthy matched control participants administered a single 300 mg oral tablet of vaniprevir
- Healthy Control for Severe HI: Healthy matched control participants administered a single 200 mg oral tablet of vaniprevir
Period: Overall Study
Arm/Group | Mild Hepatic Insufficiency (HI) | Healthy Control for Mild HI | Moderate HI | Healthy Control for Moderate HI | Severe HI | Healthy Control for Severe HI
Started | 10 | 10 | 10 | 10 | 10 | 10
Completed | 10 | 10 | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mild Hepatic Insufficiency (HI) | Healthy Control for Mild HI | Moderate HI | Healthy Control for Moderate HI | Severe HI | Healthy Control for Severe HI | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.3 (5.03) | 52.1 (3.54) | 52.1 (6.51) | 53.3 (4.90) | 53.4 (6.08) | 52.6 (7.04) | 52.3 (5.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 1 | 4 | 4 | 14
  Male | 8 | 8 | 9 | 9 | 6 | 6 | 46

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) (0-infinity) of Vaniprevir in Blood Plasma Following Single Dose Administration
Description: Participants were administered a single dose of vaniprevir; then their blood was collected at the following time points: 0.5, 1, 1.5, 2, 3, 4, 8, 12, 16, 24, 32 and 48 hours postdose. The AUC (0-infinity) of vaniprevir in blood plasma was based on an analysis of covariance (ANCOVA) model used to analyze natural log-transformed values that were back-transformed to derive geometric least-squares mean and confidence interval.
Time Frame: 0-48 hours postdose
Population: Participants administered at least one dose of investigational drug. AUC for one participant with Mild HI was not estimated due to poor correlation of the linear regression.
Measure: Geometric Mean (95% Confidence Interval); unit: µM.hr
Arm/Group | Mild Hepatic Insufficiency (HI) | Healthy Control for Mild HI | Moderate HI | Healthy Control for Moderate HI | Severe HI | Healthy Control for Severe HI
Number analyzed (Participants) | 9 | 10 | 10 | 10 | 10 | 10
µM.hr | 2.68 [1.39 to 5.18] | 1.48 [0.84 to 2.59] | 5.09 [2.21 to 11.70] | 1.64 [0.67 to 3.98] | 7.79 [5.03 to 12.00] | 0.925 [0.61 to 1.41]
Statistical Analysis 1: Comparison: Mild Hepatic Insufficiency (HI) vs Healthy Control for Mild HI; Test type: Non-Inferiority or Equivalence — If the 90% Confidence Interval falls within the interval [0.50, 2.00], then treatment of HI participants is similar to treatment of healthy matched for mild HI participants; Geometric Least-Square Mean Ratio = 1.82, 90% CI 2-sided [0.96 to 3.43]
Statistical Analysis 2: Comparison: Moderate HI vs Healthy Control for Moderate HI; Test type: Non-Inferiority or Equivalence — If the 90% Confidence Interval falls within the interval [0.50, 2.00], then treatment of HI participants is similar to treatment of healthy matched for moderate HI participants; Geometric Least-Square Mean Ratio = 3.11, 90% CI 2-sided [1.60 to 6.04]
Statistical Analysis 3: Comparison: Severe HI vs Healthy Control for Severe HI; Test type: Non-Inferiority or Equivalence — If the 90% Confidence Interval falls within the interval [0.50, 2.00], then treatment of HI participants is similar to treatment of healthy matched for severe HI participants; Geometric Least-Square Mean Ratio = 8.42, 90% CI 2-sided [5.20 to 13.64]

2. Secondary Outcome: Maximum Concentration (Cmax) of Vaniprevir in Blood Plasma Following Single Dose Administration
Description: Participants were administered a single dose of vaniprevir; then their blood was collected at the following time points: 0.5, 1, 1.5, 2, 3, 4, 8, 12, 16, 24, 32 and 48 hours postdose. The Cmax of vaniprevir in blood plasma was based on an ANCOVA model used to analyze natural log-transformed values that were back-transformed to derive geometric least-squares mean and confidence interval.
Time Frame: 0-48 hours postdose
Population: Participants administered at least one dose of investigational drug.
Measure: Geometric Mean (95% Confidence Interval); unit: µM
Arm/Group | Mild Hepatic Insufficiency (HI) | Healthy Control for Mild HI | Moderate HI | Healthy Control for Moderate HI | Severe HI | Healthy Control for Severe HI
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
µM | 0.922 [0.44 to 1.94] | 0.586 [0.29 to 1.17] | 1.88 [0.88 to 4.01] | 0.852 [0.38 to 1.91] | 2.06 [1.37 to 3.12] | 0.335 [0.23 to 0.50]
Statistical Analysis 1: Comparison: Mild Hepatic Insufficiency (HI) vs Healthy Control for Mild HI; Test type: Superiority or Other; Geometric Least-Square Mean Ratio = 1.57, 90% CI 2-sided [0.76 to 3.24]
Statistical Analysis 2: Comparison: Moderate HI vs Healthy Control for Moderate HI; Test type: Superiority or Other; Geometric Least-Square Mean Ratio = 2.21, 90% CI 2-sided [1.21 to 4.03]
Statistical Analysis 3: Comparison: Severe HI vs Healthy Control for Severe HI; Test type: Superiority or Other; Geometric Least-Square Mean Ratio = 6.16, 90% CI 2-sided [3.90 to 9.71]

ADVERSE EVENTS:
Time Frame: Up to 14 days after administration of study drug
Arm/Group | Mild Hepatic Insufficiency (HI) | Healthy Control for Mild HI | Moderate HI | Healthy Control for Moderate HI | Severe HI | Healthy Control for Severe HI
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 2/10 | 1/10 | 1/10 | 2/10 | 0/10 | 0/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mild Hepatic Insufficiency (HI) (N=10) | Healthy Control for Mild HI (N=10) | Moderate HI (N=10) | Healthy Control for Moderate HI (N=10) | Severe HI (N=10) | Healthy Control for Severe HI (N=10)
Hypersplenism (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.